CLINICAL TRIAL: NCT04217499
Title: Pelvic Ring Fractures: New Analysis Method and Treatment Decision Algorithm
Acronym: BASSINJO
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BASSINJO
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pelvic ring fractures: This retrospective study will be carried out on the data of patients who have received treatment or followed for a pelvic ring fracture, in the Orthopedic Surgery department of the Paris Saint-Joseph Hospital Group between January 2015 and September 2019.

SUMMARY:
Pelvic ring fractures are common and often the result of high energy trauma but also sometimes of lower energy trauma in older patients. A good classification and description of the fracture is essential to the choice of treatment.

The classifications used to describe these fractures are numerous (Tile modified AO, Young and Burgess, Letournel, Rommens) and of a descriptive order more or less depending on the lesion mechanism allowing some to orient the surgical reduction technique. However, none of them helps with the choice of surgical or functional treatment, which is currently based on obvious notions of instability and / or displacement of lesions and, by habit, all different services.

In addition, the complexity of these classifications leads to poor reproducibility of these.

A new method for analyzing unitary lesions has been developed in the Orthopedic Surgery department of the Paris Saint-Joseph Hospital Group with a rating system which determines the indication according to the score.

Teaching this new method of analyzing pelvic ring fractures would simplify decision making between surgical and functional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged> 18 years
* Patient treated or followed within the Orthopedic Surgery service of the GHPSJ for a pelvic ring fracture
* complete initial imaging patient record (scanner)
* French speaking patient

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients objecting to the use of their data for this research
* Patient with isolated sacral or acetabular fracture
* Absence of scanner during the initial assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were hospitalized or consulted in the Orthopedic Surgery service of the Paris Saint-Joseph Hospital Group, for the management of a pelvic ring fracture from January 2015 until September 2019.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
State of play of the decision for surgical sanction of pelvic ring fractures | Day 1
  This corresponds to the number of patients for whom surgical decisions have been made.

SECONDARY OUTCOMES:
Impact of the teaching of the new method of analysis on the surgical decision within each group | Day 1
  This corresponds to the number of files for which surgical decision-making was modified before and after teaching of the new method of analysis.
Reproducibility of this intra and inter-group decision before and after teaching | Day 1
  This corresponds to the number of files for which surgical decision-making was modified before and after teaching of the new method of analysis in intra and inter-group.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume RIOUALLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France